CLINICAL TRIAL: NCT03768076
Title: Parosteal OsTeosarcoma: a Single Istitution Experience
Brief Title: an Istitution Experience on Parosteal OsTeosarcoma
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: POsT
Record Dates: First submitted 2018-11-22; First posted 2018-12-07 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Parosteal Osteosarcoma
MeSH Terms: conditions — Osteosarcoma, Juxtacortical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
single institution cases series review of histological and clinical data

DETAILED DESCRIPTION:
Investigators will review all the cases with a diagnosis of primary parosteal osteosarcoma treated at the Rizzoli Institute from 1900 up to 31 July 2018, retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Institute from 01 Jan 1900 to 31 Jul 2018
* Diagnosis of parosteal osteosarcoma
* Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

• Patients with histological diagnosis different from parosteal osteosarcoma

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: male and female with diagnosis of parosteal osteosarcoma treated at Rizzoli institute from 01 Jan 1900 to 31 Jul 2018
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
retrospective analysis of cases of Parosteal osteosarcoma | at baseline (Day0)
  Investigators will exam the presence of progression (dedifferentiation) areas and the relationship of these factors to individual outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
No Individual Patient Data sharing plan has been implemented

REFERENCES:
- [Result] Han I, Oh JH, Na YG, Moon KC, Kim HS. Clinical outcome of parosteal osteosarcoma. J Surg Oncol. 2008 Feb 1;97(2):146-9. doi: 10.1002/jso.20902. PMID 18050289
- [Result] Bertoni F, Bacchini P, Staals EL, Davidovitz P. Dedifferentiated parosteal osteosarcoma: the experience of the Rizzoli Institute. Cancer. 2005 Jun 1;103(11):2373-82. doi: 10.1002/cncr.21039. PMID 15852358
- [Result] Okada K, Frassica FJ, Sim FH, Beabout JW, Bond JR, Unni KK. Parosteal osteosarcoma. A clinicopathological study. J Bone Joint Surg Am. 1994 Mar;76(3):366-78. doi: 10.2106/00004623-199403000-00007. PMID 8126042
- [Result] Laitinen M, Parry M, Albergo JI, Jeys L, Abudu A, Carter S, Sumathi V, Grimer R. The prognostic and therapeutic factors which influence the oncological outcome of parosteal osteosarcoma. Bone Joint J. 2015 Dec;97-B(12):1698-703. doi: 10.1302/0301-620X.97B12.35749. PMID 26637687

DOCUMENTS (1):
  • Study Protocol (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT03768076/Prot_000.pdf